CLINICAL TRIAL: NCT05193409
Title: A Phase 2, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of BNC210 Compared to Placebo for the Acute Treatment of Social Anxiety Disorder
Brief Title: A Phase 2 Study of BNC210 for the Acute Treatment of Social Anxiety Disorder
Acronym: PREVAIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionomics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNC210.013
Record Dates: First submitted 2022-01-03; First posted 2022-01-14 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 225 mg BNC210 (Experimental)
  Interventions: Drug: 225 mg BNC210
- 675 mg BNC210 (Experimental)
  Interventions: Drug: 675 mg BNC210
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 225 mg BNC210 — 225 mg BNC210
  Arms: 225 mg BNC210
Drug: 675 mg BNC210 — 675 mg BNC210
  Arms: 675 mg BNC210
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of an acute dose of BNC210 compared to placebo on reducing anxiety provoked by a speaking challenge and measured using the Subjective Units of Distress Scale (SUDS) in patients with Social Anxiety Disorder (SAD).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 3-arm, parallel-group, multi-center study. Participants will attend a Screening Visit to confirm eligibility and then return to the clinic within 14 days to be randomized into the study. Randomized participants will receive a single dose of their allocated study intervention (225 mg BNC210, 675 mg BNC210 or placebo) and approximately 1 hour later participate in a speaking challenge. After 1 week, a safety follow-up assessment will be conducted by phone/video conference.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a current diagnosis of Social Anxiety Disorder (SAD) as defined in DSM-5 and confirmed by Structured Clinical Interview for DSM-5 Disorders - Clinical Trials version (SCID-5-CT).
* Liebowitz Social Anxiety Scale (LSAS) total score of ≥70
* Suitable contraception use in line with protocol requirements
* Ability to swallow tablets

Exclusion Criteria:

* History of schizophrenia, bipolar disorder, or psychotic disorders, or has a current clinically predominant diagnosis of any other Axis I disorder, other than SAD
* Hamilton Rating Scale for Depression (HAM-D) score of ≥18
* Moderate or severe alcohol-use disorder, or any other substance-use disorder (any severity) in the past 12 months
* Use of psychotropic medications within 30 days of screening. Daily use of benzodiazepines within 90 days of screening.
* Previous participation in a study that involved a speaking challenge.
* Any clinically significant medical history or findings as determined by the Investigator that could interfere with the objectives of the study or put the participant at risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - PREVAIL Study Clinical Trial Site, Beverly Hills, California
  - PREVAIL Study Clinical Trial Site, Encino, California
  - PREVAIL Study Clinical Trial Site, Glendale, California
  - PREVAIL Study Clinical Trial Site, New Haven, Connecticut
  - PREVAIL Study Clinical Trial Site, Lauderhill, Florida
  - PREVAIL Study Clinical Trial Site, Miami, Florida
  - PREVAIL Study Clinical Trial Site, Miami Lakes, Florida
  - PREVAIL Study Clinical Trial Site, Decatur, Georgia
  - PREVAIL Study Clinical Trial Site, Prairie Village, Kansas
  - PREVAIL Study Clinical Trial Site, Boston, Massachusetts
  - PREVAIL Study Clinical Trial Site, Princeton, New Jersey
  - PREVAIL Study Clinical Trial Site, Brooklyn, New York
  - PREVAIL Study Clinical Trial Site, Charlotte, North Carolina
  - PREVAIL Study Clinical Trial Site, Cincinnati, Ohio
  - PREVAIL Study Clinical Trial Site, Draper, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Papapetropoulos S, Doolin E, Odontiadis M, Paul D, Jaros M, Rolan P, Taylor C, Stein MB. A phase 2, placebo-controlled study to evaluate the efficacy and safety of BNC210, an alpha-7 nicotinic receptor negative allosteric modulator, for acute, as-needed treatment of social anxiety disorder (SAD) - The PREVAIL study. Psychiatry Res. 2025 Apr;346:116387. doi: 10.1016/j.psychres.2025.116387. Epub 2025 Feb 10. PMID 39954310

RESULTS

PARTICIPANT FLOW:
Groups:
- 225 mg BNC210: 225 mg BNC210 tablet single dose
- 675 mg BNC210: 675 mg BNC210 tablet single dose
- Placebo: Placebo tablet single dose
Period: Overall Study
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo
Started | 50 | 51 | 50
Completed | 50 | 51 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo | Total
Number analyzed (Participants) | 50 | 51 | 50 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (11.55) | 37.7 (12.86) | 34.5 (9.49) | 35.9 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 27 | 95
  Male | 17 | 16 | 23 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 12 | 43
  Not Hispanic or Latino | 35 | 35 | 38 | 108
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 7 | 7 | 9 | 23
  White | 39 | 40 | 36 | 115
  More than one race | 2 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Liebowitz Social Anxiety Scale (LSAS) [Mean (Standard Deviation); unit: units on a scale] — The Liebowitz Social Anxiety Scale (LSAS) is a clinician administered rating scale used for the quantification of symptomatic distress and impairment caused by social anxiety disorder (SAD). The scale includes 24 items divided into two subscales (fear or anxiety, and avoidance) that evaluate social, interactional and performance situations. Scores on each of the items are added to give a global score ranging from 0-144, with higher scores indicating greater severity of SAD symptoms.
  units on a scale | 98.7 (15.75) | 98.3 (16.98) | 95.3 (16.34) | 97.4 (16.33)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Average Subjective Units of Distress Scale (SUDS) Score of the 5-minute Performance Phase of a Public Speaking Challenge
Description: The SUDS is a self reported measure of the intensity of distress currently experienced by an individual. The range is 0-100, with a higher score indicating a higher level of anxiety/greater distress.
Time Frame: Assessed over a single visit: Baseline; and the Performance Phase (0,1,2,3,4,5 minutes) of the Public Speaking Challenge, conducted 1 hour post-dose.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo
Number analyzed (Participants) | 50 | 51 | 50
score on a scale | 22.42 [15.78 to 29.06] | 24.26 [17.70 to 30.82] | 29.03 [22.44 to 35.62]

2. Secondary Outcome: Change From Baseline to the Average SUDS Score of the 2-minute Anticipation Phase of a Public Speaking Challenge
Description: as for outcome 1
Time Frame: Assessed over a single visit: Baseline; and the Anticipation Phase (0,1,2 minutes) of the Public Speaking Challenge, conducted 1 hour post-dose.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo
Number analyzed (Participants) | 50 | 51 | 50
score on a scale | 15.18 [9.57 to 20.79] | 12.86 [7.31 to 18.41] | 18.95 [13.37 to 24.52]

3. Secondary Outcome: Change From Baseline to the End of the 5-minute Performance Phase of Public Speaking Challenge in the State-Trait Anxiety Inventory (State Component; STAI-State) Score
Description: The STAI-State is a self reported measure of subjective anxiety at the time of questionnaire completion. The range is 0-80 with a higher total score indicating a higher level of anxiety.
Time Frame: Assessed over a single visit: Baseline; and the Performance Phase (5 minutes) of the Public Speaking Challenge, conducted 1 hour post-dose.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo
Number analyzed (Participants) | 50 | 51 | 50
score on a scale | 3.83 [0.17 to 7.50] | 3.04 [-0.06 to 6.69] | 4.71 [1.04 to 8.39]

4. Secondary Outcome: Change From Baseline to the End of the 2-minute Anticipation Phase of Public Speaking Challenge in the STAI-State Score
Description: as for outcome 3
Time Frame: Assessed over a single visit: Baseline; and the Anticipation Phase (2 minutes) of the Public Speaking Challenge, conducted 1 hour post-dose.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo
Number analyzed (Participants) | 50 | 51 | 50
score on a scale | 5.77 [2.77 to 8.78] | 5.45 [2.47 to 8.43] | 9.04 [6.04 to 12.04]

5. Secondary Outcome: Change From Baseline to the End of the 5-minute Performance Phase of Public Speaking Challenge in the Self Statements During Public Speaking - Negative Self Statements (SSPS-N) Score
Description: The SSPS-N is a self reported measure that assesses cognitions related to public speaking.The range is 0-25 with a higher total score indicating a higher level of negative cognitions.
Time Frame: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo
Number analyzed (Participants) | 50 | 51 | 50
score on a scale | -1.54 [-3.07 to -0.01] | -1.79 [-3.34 to -0.24] | -0.77 [-2.29 to 0.75]

6. Secondary Outcome: Change From Baseline to the End of the 2-minute Anticipation Phase of Public Speaking Challenge in the SSPS-N Score
Description: as for outcome 5
Time Frame: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo
Number analyzed (Participants) | 50 | 51 | 50
score on a scale | -0.38 [-1.72 to 0.97] | -2.69 [-4.05 to -1.33] | -1.25 [-2.58 to 0.08]

7. Post Hoc Outcome: Change From Baseline in the Area Under the Curve (AUC) of the Combined SUDS Scores of the Anticipation and Performance Phases of a Public Speaking Challenge.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: To increase the sample size for the post-hoc analysis, data were combined for the two active BNC210 treatment groups versus placebo. Only participants who completed the public speaking challenge were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale * minutes
Groups:
- 225 mg BNC210 and 675 mg BNC210: Participants from both active BNC210 treatment groups
Arm/Group | 225 mg BNC210 and 675 mg BNC210 | Placebo
Number analyzed (Participants) | 85 | 47
score on a scale * minutes | 229.1 [170.7 to 287.4] | 325.9 [250.4 to 401.4]

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- 225 mg BNC210: 225 mg BNC210 single dose
- 675 mg BNC210: 675 mg BNC210 single dose
- Placebo: Placebo single dose
Arm/Group | 225 mg BNC210 | 675 mg BNC210 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 6/50 | 10/51 | 3/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 225 mg BNC210 (N=50) | 675 mg BNC210 (N=51) | Placebo (N=50)
Somnolence (Nervous system disorders) | 2 | 6 | 2
Headache (Nervous system disorders) | 3 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT05193409/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT05193409/SAP_001.pdf